CLINICAL TRIAL: NCT02037061
Title: A Randomized Control Trial on the Effect of Local Analgesia on Postoperative Gluteal Pain in Patients Undergoing Sacrospinous Ligament Colpopexy
Brief Title: Reducing Post-Op Pain After Sacrospinous Ligament Colpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1413
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Placebo Comparator): Intraoperatively the patient will receive 10ml of normal saline injected into the sacrospinous ligament.
  Interventions: Other: Normal Saline
- bupivacaine (Active Comparator): Intraoperatively the patient will receive 10 ml of bupivacaine injected into the sacrospinous ligament.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Intraoperatively the patient will receive 10ml of bupivacaine injected into the sacrospinous ligament.
  Arms: bupivacaine
Other: Normal Saline
  Arms: normal saline

SUMMARY:
This is a randomized controlled trial to determine if intraoperative local analgesia administered at the level of the sacrospinous ligament can lessen the gluteal pain felt by patients postoperatively after SSL colpopexy.

Hypothesis: Local analgesia administered at the level of the sacrospinous ligament can lessen the gluteal pain felt by patients postoperatively after SSL colpopexy.

DETAILED DESCRIPTION:
This is a randomized double-blind clinical trial. Potential subjects will be identified by members of the Center for Urogynecology and Pelvic Reconstructive Surgery at the Cleveland Clinic main campus. Eligible patients that agree to participate will be provided written informed consent administered by the collaborators listed on the IRB at the Cleveland Clinic main campus.

All subjects will be predetermined by their surgeon to undergo sacrospinous ligament colpopexy for management of vaginal apex prolapse after hysterectomy. The participants will then be randomized to one of two groups: "local analgesia injection" or "normal saline injection" according to a computer-generated randomization schedule with random block sizes with the use of the SAS statistical software package (SAS Institute, Cary, NC). Randomization will be done by a nurse coordinator who will not be involved in participant recruitment or injection at the time of surgery. All patients and providers will be blinded to their assignment. The assignment will be kept in an envelope which will be given to the pharmacy the day of the patient's scheduled procedure. The pharmacy will then dispense the correct intervention based on the randomization.

In addition to a standardized evaluation including the history and physical examination, patients will be asked to complete a functional assessment questionnaire as well as a surgical pain scale at the preoperative visit. Prior to discharge from the hospital, patients will be provided with an envelope with pre-labeled questionnaires to bring home with them. Prior to discharge, they will be asked to complete the surgical pain scale only. Subjects will then be called the day after discharge, at week 1, week 2, week 4 and week 6 after the procedure and will be reminded to complete the appropriate questionnaires/forms that were provided to them. They will bring in these forms to their 6-week postoperative visit. All questionnaires will be self-administered. Completion of these questionnaires is the only additional assessment that is specific to participation in this study and is not usually included as part of the standard care of sacrospinous ligament colpopexy.

Sacrospinous ligament colpopexy will be performed in a standard fashion. The approach is done by either entering the vagina along the anterior or posterior wall or at the apex. Approach and side of the suspension will be based on surgeon's preference. Prior to entry, the apex of the vaginal vault is first identified by visualizing the old hysterectomy scar. Allis clamps are used to demarcate the new vaginal apex and to ensure that this apex will suspend adequately to the sacrospinous ligament, which is identified transvaginally by palpation of the ischial spine. Once vaginal entry is made, sharp and blunt dissection are performed down to the pararectal space on one or both sides. Identification of the ischial spine confirms the position of the coccygeus-sacrospinous ligament complex. Once the complex is freed of any overlying areolar tissue, a Briesky Navratil retractor is placed to retract the rectum away from the site of suture placement and to help with visualization of the ligament complex.

The CapioTM device is then used to place the suspension sutures. 3 sutures are placed: 2 delayed-absorbable (0 PDS) and 1 permanent (0 prolene). All sutures are placed one and a half to two fingerbreadths (2-3cm) medial to the ischial spine in a sequential fashion. After placement, a rectal exam is done to ensure that no sutures have been placed through the rectum and the coccygeus-sacrospinous ligament complex is visualized carefully to ensure that the surgical site is hemostatic. The absorbable-delayed suspension sutures are placed through the vaginal epithelium at the level of the neoapex and all permanent sutures are placed through the subepithelial tissue.

Injection of the sacrospinous ligament will be performed prior to tying down the suspension sutures according to the group the patient is randomized to. A pudendal nerve block kit needle and syringe will be used to administer the injection. The spacer will be removed, allowing the needle point to enter the ligament 10mm in depth with each injection. The injection will be placed in 3 locations (~3mL in each injection for a total of 10mL) along the center of the sacropinous ligament under each previously placed suture. Proper injection technique will be performed with each injection (e.g. there will be confirmation of extravascular placement of the needle tip prior to each injection). One of two injections (bupivacaine vs. normal saline) delivered by the pharmacy will be administered depending upon the group to which the patient has been randomized.

Preoperative data will include the following:

* Patient age, race, vaginal parity, menopausal sate, tobacco use, BMI, prior prolapse surgery, preoperative prolapse stage (see Appendix for demographic data sheet)
* Assessment of functional status, surgical pain scale
* Labs (Hb/Hct)

Intraoperative data will include the following:

* Surgery date
* Surgeon
* Side of Colpopexy
* Concomitant procedures
* EBL

Postoperative data will include the following:

* Days in the hospital
* Pain medication requirment during hospitalization
* Prior to discharge from hospital: surgical pain scale; localization of pain
* POD#1: Labs (Hb/Hct)
* Time from surgery [incision] to discharge (hours)
* 1st postoperative week oDaily surgical pain scale with localization of pain oDaily pain medication use oAt end of week 1: Assessment of functional status
* 2nd postoperative week oDaily surgical pain scale with localization of pain oDaily pain medication use oAt end of week 2: Assessment of functional status
* 4th postoperative week (at end of week 4) oAssessment of functional status oSurgical pain scale with localization of pain
* 6th postoperative week (at end of week 6) oAssessment of functional status oSurgical pain scale with localization of pain
* Date of 6-week postoperative
* Need for intervention for pain: trigger point injection, PFPT referral, reoperation

All paper forms used for data collection will be kept in a research cabinet dedicated to this project which will be locked at all times, in a locked office at the Cleveland Clinic. All forms will contain de-identified information - identification numbers will correspond to the subjects listed in the master excel file.

All study data will be transferred and managed electronically using REDCap (Research Electronic Data Capture). Each subject will be entered into REDCap using the assigned identification number from the master excel file. REDCap is a secure, web-based application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation, audit trials, and a de-identified data export mechanism to common statistical packages. They system was developed by a multi-institutional consortium which was initiated at Vanderbilt University and includes the Cleveland Clinic. The database is hosted at the Cleveland Clinic Research Datacenter in the JJN basement and is managed by the Quantitative Health Sciences Department. The system is protected by a login and Secure Sockets Layers (SSL) encryption. Data collection is customized for each study as based on a study-specific data dictionary defined by the research team with guidance from the REDCap administrator in Quantitative Health Sciences at the Cleveland Clinic

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, who are to undergo sacrospinous ligament colpopexy for vaginal apex prolapse after hysterectomy
* Other concomitant prolapse and anti-incontinence procedures (e.g., anterior colporrhaphy, paravaginal defect repair, posterior colporrhaphy, or mid-urethral sling procedures) will be performed at the primary surgeon's discretion

Exclusion Criteria:

* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Need for concomitant surgeries not related to pelvic organ prolapse or incontinence
* Chronic pain conditions (e.g., fibromyalgia, myositis, myofascial pain syndrome)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Unger, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrando CA, Walters MD. A randomized double-blind placebo-controlled trial on the effect of local analgesia on postoperative gluteal pain in patients undergoing sacrospinous ligament colpopexy. Am J Obstet Gynecol. 2018 Jun;218(6):599.e1-599.e8. doi: 10.1016/j.ajog.2018.03.033. Epub 2018 Mar 31. PMID 29614274

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: Intraoperatively the patient will receive 10ml of normal saline injected into the sacrospinous ligament.
  Normal Saline
Period: Overall Study
Arm/Group | Normal Saline | Bupivacaine
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Bupivacaine | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7) | 63 (9) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Gluteal Pain
Description: Pain measured using a pain numeric rating scale from 0 to 10 (0=no pain, 10= worst pain imaginable)
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Bupivacaine
Number analyzed (Participants) | 22 | 24
units on a scale
  Mean gluteal pain in immediate post op | 3.6 (2.7) | 4.0 (2.9)
  Mean gluteal pain within week 1 of procedure | 2.0 (2.4) | 2.0 (2.6)
  Mean gluteal pain 2 weeks after procedure | 1.1 (1.3) | 1.0 (1.1)
  Mean gluteal pain 4 weeks after procedure | 0.3 (0.5) | 0.3 (0.4)
  Mean gluteal pain 6 weeks after procedure | 0.1 (0.3) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Normal Saline vs Bupivacaine; Test type: Other; p = 0.83, t-test, 2 sided

2. Secondary Outcome: Need for Intervention for Postoperative Pain
Description: Need for intervention through the use of trigger point injection, referral to pelvic floor physical therapy, or reoperation
Time Frame: 6-weeks
Measure: Number; unit: participants
Arm/Group | Normal Saline | Bupivicaine
Number analyzed (Participants) | 22 | 24
participants
  Trigger point injection | 0 | 0
  Referral to pelvic floor physical therapy | 0 | 0
  Reoperation | 0 | 0

3. Secondary Outcome: Overall Pain Beyond Day of Discharge
Description: Pain measured using the pain numeric rating scale from 0-10 (0=no pain, 10= worst pain imaginable)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Bupivicaine
Number analyzed (Participants) | 22 | 24
units on a scale
  Mean overall pain 2 weeks after procedure | 1.1 (0.3) | 1.0 (0.2)
  Mean overall pain 4 weeks after procedure | 0.3 (0.1) | 0.3 (0.1)
  Mean overall pain 6 weeks after procedure | 0.1 (0.1) | 0.1 (0.1)

ADVERSE EVENTS:
Arm/Group | Normal Saline | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes